CLINICAL TRIAL: NCT05852301
Title: Optimising Cohorts for HIV Cure Interventions: the Role of Very High CD4 T Cell Counts: HI-ART Study
Brief Title: Optimising Cohorts for HIV Cure Interventions
Acronym: HI-ART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: The Peter Doherty Institute for Infection and Immunity (Other)
Responsible Party: Sponsor
Other Study IDs: 413.22
Record Dates: First submitted 2023-04-17; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-04

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- HI-ART: People living with HIV with CD4+ T cells > 800 c/uL on ART initiation
  Interventions: Other: no intervention
- HI-ART control: People living with HIV with CD4+ T cells between 500-800 c/uL on ART initiation
  Interventions: Other: no intervention
- Hyper: People living with HIV with CD4+ T cells >800 c/μL on ART initiation, but increase to >1000c/μL within 48 months of ART initiation
  Interventions: Other: no intervention
- Hyper control: People living with HIV with CD4+ T cells <500 c/μL on ART initiation and reconstituted to 500-1000c/μL within 48 months of ART initiation
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention, observational study only

SUMMARY:
In a recent international substudy of START (Study of Initiation of ART in Early HIV Infection), we found that people with HIV (PHIV) who initiate ART with CD4+ T cells > 800 cells/μL achieve a substantially smaller HIV reservoir on ART, as measured by the frequency of CD4+ T cells containing HIV DNA, compared to individuals who commence ART with CD4 counts between 500-599 and 600-799 cells/µL. We have termed these individuals 'HI-ARTs' (very High CD4 prior to ART).

Smaller reservoirs have also been noted in PHIV who achieve a CD4 count greater than 1000 cells/µL within 48 months of initiation of ART who are referred to as 'Hypers'.

This study will establish a prospective cohort of HI-ARTs and Hypers at Alfred Health and our clinical partners. It will characterise the HIV reservoir and HIV-specific immune responses in these individuals and compare these to age-matched HIV positive controls from the Alfred HIV clinic, who have CD4+ T cells between 500-800 cells/uL, or who do not reconstitute their CD4+ T cells to greater than 1000 cells/uL within 48 months.

Participants will be asked to donate a blood sample at baseline, and pending initial analyses, again at month 12 and 24.

DETAILED DESCRIPTION:
In individuals who commence ART in early HIV infection (within 6 months of acquiring HIV) compared to those who initiate ART in later infection, the frequency of cells containing intact and replication competent HIV DNA is reduced and HIV-specific immune responses are better preserved.

Previous studies in humans and infected macaque models have demonstrated that smaller reservoirs (measured by HIV DNA levels) predicted a longer time to viral rebound when ART was interrupted. These individuals are difficult to identify, and specialist research laboratories are required to conduct HIV DNA assays. There is therefore an urgent need to develop simple and efficient processes to identify PHIV with small HIV reservoirs who may best respond to cure interventions aiming to control virus without the need for regular ART.

In a recent international substudy of the START study (Initiation of ART in Early HIV Infection), our group showed that PHIV who initiate ART with CD4 T cells > 800 cells/μL achieve a substantially smaller HIV reservoir on ART compared to individuals who commence ART with CD4 counts between 500-800 cells/μL. We have termed these individuals 'Hi-ARTs' (High CD4 prior to ART). Smaller reservoirs have also been noted in PHIV who reach a CD4 count above 1000 cells/μL within 48 months of ART initiation who are referred to as 'Hypers'.

The immunological mechanisms by which latently infected cells are more efficiently eliminated or diluted by uninfected CD4 T cells in these patient groups are not understood. It is also unclear whether cells containing genetically-intact (or replication competent) HIV are eliminated at the same rate as cells harbouring HIV with extensive mutations/deletions ('defective'). The distinction between cells harbouring intact or defective HIV is important as only intact virus can cause viral rebound in the absence of ART and there are now assays to distinguish between the two.

Blood on enrolment and yearly for 2 years. Plasma and peripheral blood mononuclear cells (PBMC) will be assessed to determine the reservoir size and HIV-specific immune responses using validated assays including total HIV DNA and Intact Proviral DNA (IPDA), cell associated unspliced HIV-RNA (transcriptional activity), plasma HIV RNA, and intracellular cytokine staining in response to Gag and Nef stimulation using antibodies against IFN-g, TNF-a, and CD107a. Outcome measures will be compared and age- and sex- matched controls from The Alfred Hospital HIV clinic.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Able to give written informed consent;
* Documented HIV infection (antibody positive);
* Taking continuous ART for at least 2 years prior to study enrolment;

Exclusion Criteria:

* Unwillingness to follow protocol requirements;
* HIV negative;
* Not meeting study definition for HI-ART or Hyper (except for control group);
* Medicare ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who are HIV antibody positive; have very high CD4 counts on ART initiation (>800 cells/uL , known as HI-ARTs), or reconstitute their CD4 counts to >1000 cells/μL within 48 months of commencing ART (Hypers) will be eligible for inclusion.
  The study will recruit people with HIV into 4 cohorts based on CD4+ T cell criteria.
  * CD4+ T cells > 800 c/uL on ART initiation (HI-ARTs)
  * CD4+ T cells between 350-800 c/uL on ART initiation (HI-ART controls)
  * CD4+ T cells <800 c/μL on ART initiation, but increase to >1000c/μL within 48 months of ART initiation (Hypers)
  * CD4+ T cells reconstituted to 500-1000c/μL within 48 months (Hyper controls)
  The study consists of three study visits over 24 months with study visits and blood sampling at months 0, 12 and 24.
Sampling Method: Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
HIV-DNA | at baseline
  Quantitative DNA measurements in CD4+ T cells by PCR

SECONDARY OUTCOMES:
Reservoir measurements | at baseline
  Quantitative HIV RNA/DNA measurements in CD4+ T cells by PCR
Reservoir measurements | at baseline
  flow cytometry
Reservoir measurements | at baseline
  proviral sequencing
HIV-specific T-cell responses | at baseline
  HIV-specific T-cell immunity by intracellular cytokine staining (ICS) to measure the frequency of responding cells producing multiple effector cytokines including IFN-γ, TNF-α, and IL-2.
Decay of reservoir | at 12 months
  Compare changes in intact/defective HIV DNA by PCR from baseline
Decay of reservoir | at 24 months
  Compare changes in intact/defective HIV DNA by PCR from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Lau, MBBS, Principal Investigator — The Alfred
Locations (1):
- Alfred Health, Prahran, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided